CLINICAL TRIAL: NCT06817967
Title: A Prospective, Randomised, Double-blind, Multicentre Parallel-group Study Comparing a Medical Device: Proponent Solution - Nasal Spray (PSNS) With Comparator (Sodium Chloride 0.9%) for Treatment of Nasal Congestion Symptoms (in Adults) During Rhinitis Medicamentosa While Weaning From Direct-acting Alpha-adrenergic Agonists, Such as Xylometazoline or Oxymetazoline
Brief Title: A Study Comparing Proponent Solution - Nasal Spray (PSNS) With Salt Water for Treating Nasal Congestion Symptoms in Adults With Rebound Nasal Congestion While Weaning From Nasal Decongestant Sprays
Acronym: PROUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharma Nordic AS (Industry)
Collaborators: Proponent Biotech GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROUD study
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-02

CONDITIONS: Rhinitis Medicamentosa

STUDY DESIGN:
Intervention Model Description: This was a prospective, randomised, double-blind, multicentre, parallel-group study to evaluate Proponent Solution - Nasal Spray (PSNS) compared to Isotonic Saline Nasal Spray (ISNS) for treatment of nasal congestion symptoms in adult subjects with RM while weaning from direct-acting alpha-adrenergic agonists, such as xylometazoline or oxymetazoline. The study aimed to recruit approximately 200 subjects (actual: 194 subjects) who should receive 4-weeks (28 days, 1 to +5 days) of treatment with PSNS or ISNS, to evaluate the efficacy, safety, and tolerability.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects were randomly assigned to treatment with PSNS or ISNS using a block size of 4. Randomisation codes were assigned strictly sequentially as subjects were eligible for randomisation. The randomisation list was generated by an independent statistician and was kept strictly confidential. The investigational medicinal device and the comparator nasal spray were distributed in identical packages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PSNS (Experimental): The PSNS consisted of a Locke-Ringer solution containing 10 mg/mL sodium propionate. The solution was provided in a microbiologically safeguarded, multi-use dosing system consisting of a plastic storage bottle (20 mL) and a nasal applicator. The nasal spray was self-administered by study subjects at a maximum daily dose of 16 puffs per day, distributed over 1-2 puffs per nostril 2-4 times per day, depending on symptom severity and their alleviation. Each puff contained approximately 140 µl nasal spray solution.
  Interventions: Device: PSNS
- ISNS (Placebo Comparator): The comparator ISNS consisted of water containing 0.9% w/v sodium chloride. The ISNS solution was provided in the same microbiologically safeguarded, multi-use dosing system as the investigational device product. The nasal spray was self-administered by study subjects at a maximum daily dose of 16 puffs per day, distributed over 1-2 puffs per nostril 2-4 times per day, depending on symptom severity and their alleviation. Each puff contained approximately 140 µl nasal spray solution.
  Interventions: Device: ISNS

INTERVENTIONS:
Device: PSNS — The nasal spray was self-administered by study subjects at a maximum daily dose of 16 puffs per day, distributed over 1-2 puffs per nostril 2-4 times per day, depending on symptom severity and their alleviation.
  Arms: PSNS
Device: ISNS — The nasal spray was self-administered by study subjects at a maximum daily dose of 16 puffs per day, distributed over 1-2 puffs per nostril 2-4 times per day, depending on symptom severity and their alleviation.
  Arms: ISNS

SUMMARY:
The purpose of the study was to test if the PROPONENT® nasal spray works, if it is safe, and if it helps participants to stop using addictive nasal decongestant sprays. To be able to take part in the study, participants had to be at least 18 years old, suffer from a condition called "rebound nasal congestion" or "rhinitis medicamentosa (RM)", and be dependent on nasal decongestants. Participants were randomly assigned to receive either PROPONENT® nasal spray or a nasal spray with physiological saline during the 4-week study treatment period. Neither the participants nor their doctor knew which they were receiving. In total, 194 participants took part in this study in several hospitals in Norway.

The study included three visits to the study center: one at the beginning and one at the end of the treatment period, and a follow-up visit approximately 4 weeks after the end of study treatment. During the study treatment period, participants used 1-2 puffs of study nasal spray in each nostril in the morning and evening. They could use the nasal spray additional times if they felt the need due to nasal congestion, up to a maximum of 16 puffs a day. During they study treatment period, participants were asked to measure every morning and evening how much air they could maximally inhale through their nose using a simple instrument called Peak Nasal Inspiratory Flow (PNIF) meter. At the end of each week of the treatment period, participants were asked to report how bad their nasal problems had been during the past week using electronic questionnaires. At the follow-up visit, participants were asked if they could still manage without the decongestant nasal sprays they had been using before entering the study, and if they felt that they had become addicted to the study nasal spray.

DETAILED DESCRIPTION:
This was a prospective, randomised, double-blind, multicenter, parallel-group study to evaluate Proponent Solution - Nasal Spray (PSNS) compared to sodium chloride 0.9% (Isotonic Saline Nasal Spray [ISNS]) for treatment of nasal congestion symptoms during RM while weaning from direct-acting alpha-adrenergic agonists, such as xylometazoline or oxymetazoline. The study aimed to recruit approximately 200 subjects (actual: 194 subjects) who should receive 4 weeks of treatment with PSNS or ISNS to evaluate the efficacy, safety, and tolerability.

Before study start, prospective subjects received a telephone call by the study personnel where they were informed about the study and asked to make notes of their daily use of xylometazoline or oxymetazoline each evening (including the number of doses used) for 7 days prior to start of study treatment. This data was transferred to an electronic diary (eDiary) for all subjects that were included in the study. Prospective subjects attended an enrolment visit (Visit 1) at the investigational site, where informed consent was discussed and signed. Eligible subjects were randomised (1:1) to receive the investigational device product (PSNS) or the comparator (ISNS), and self-administered the first dose of study treatment under supervision of the study personnel.

During the 4-week treatment period (28 days, -1 to +5 days), subjects self-administered the study nasal spray at a maximum dose of 16 puffs per day distributed over 1-2 puffs applied into each nostril 2-4 times daily. Subjects were asked to report daily their objective morning and evening PNIF meter results in an eDiary on a smartphone or laptop both before and 10 minutes after administration of 1-2 puffs of either PSNS or the comparator. Each week, subjects had to fill out electronic questionnaires assessing their nasal congestion/obstruction using validated scoring systems (NOSE and NOVAS-score). At 21-35 days after the end of study treatment (Visit 3), each subject was asked to complete a follow-up registration in the eDiary. During this assessment, it was also assessed whether the subject had become addicted to/physically dependent on the study nasal spray.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent prior to any study-specific procedures.
2. Be 18 years of age or older.
3. Use xylometazoline or oxymetazoline nasal spray at least once daily over a period of 7 days, registered before entering the clinical study.
4. Be diagnosed with RM by a medical doctor. The subject needed/wanted to wean from direct-acting alpha-adrenergic agonists, such as xylometazoline or oxymetazoline.

Exclusion Criteria:

1. Had influenza, acute or chronic rhinitis (other than RM), acute sinusitis, suppurative tonsillitis, pneumonia, or tuberculosis.
2. Had taken any medication or cold remedies to treat common colds (including Proponent Solution - Nasal Spray [PSNS]) within the last week.
3. Had used glucocorticoids (tablets, injections, and topical inhalers) within the last week or will need this medication during the study.
4. Had serious primary cardiovascular, kidney, liver, neurological, psychiatric, or haematological disease.
5. Had a diagnosis of asthma, chronic obstructive pulmonary disease, chronic cough, or other significant acute or chronic respiratory conditions or disorders.
6. Had an allergic disease and require daily peroral antihistamines for the treatment of the disease during the inclusion period and the study.
7. Study subject was a current smoker.
8. Nasal disorder or nasal condition as a relevant septal deviation, polyposis, chronic rhinitis, ulcer, etc., and/or reconstructive surgery, that could impair nasal breathing.
9. Had a known ongoing cancer disease.
10. Was identified by the Investigator as inappropriate to participate in this study (e.g., inability to report daily using smartphone/computer [eDiary]).
11. Participated in other clinical trials within the last 3 months.
12. Had known allergy or hypersensitivity to the components of the investigational product.
13. Were pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who did not use xylometazoline or oxymetazoline nasal spray for three consecutive days at the end of the clinical study treatment period (PSNS vs ISNS) | Day 0 (randomisation, start of treatment) until end of treatment (Day 28, -1 day until + 5 days)

SECONDARY OUTCOMES:
At least a 50% reduction in the use of xylometazoline or oxymetazoline nasal spray for three consecutive days at the end of the study treatment period compared to the use reported before study start (PSNS vs ISNS) | Day 0 (randomisation, start of treatment) until end of treatment (Day 28, -1 day until + 5 days)
  This was based on the self-reported use of xylometazoline/oxymetazoline.
Peak Nasal Inspiratory Flow (PNIF)-score measured in the last week of the study treatment period | Last week of the study treatment period (Day 27-33)
  The PNIF meter is a lightweight and compact instrument that provides an objective result of nasal patency. Study subjects were asked to take three repeated PNIF measurements at each time point, and to record the highest result in their eDiary. The PNIF score was measured in litres per minute (L/min). Values above 125 L/min were considered out-of-range. Higher values indicate better nasal patency.
NOVAS-score measured in the last week of the study treatment period | Last week of the study treatment period (Day 27-33)
  This was assessed using the validated questionnaire Nasal Obstruction Visual Analogue Scale (NOVAS). The scale ranges from 0 to 10, where 0 corresponds to "no nasal obstruction" and 10 corresponds to "maximum nasal obstruction".
NOSE-score measured in the last week of the study treatment period | Last week of the study treatment period (Day 27-33)
  This was assessed using the validated questionnaire Nasal Obstruction Symptom Evaluation (NOSE). The total score ranges from 0 to 20, and a higher score indicates more severe nasal obstruction.
Temporal trends in PNIF-score during the study treatment period | From randomisation to end of study treatment (Day 27-33)
  The PNIF meter is a lightweight and compact instrument that provides an objective result of nasal patency. Study subjects were asked to take three repeated PNIF measurements at each time point, and to record the highest result in their eDiary. The PNIF score was measured in L/min. Values above 125 L/min were considered out-of-range. Higher values indicate better nasal patency.
Temporal trends in NOVAS-score during the study treatment period | From randomisation to end of study treatment (Day 27-33)
  This was assessed using the validated questionnaire Nasal Obstruction Visual Analogue Scale (NOVAS). The scale ranges from 0 to 10, where 0 corresponds to "no nasal obstruction" and 10 corresponds to "maximum nasal obstruction".
Temporal trends in NOSE-score during the study treatment period | From randomisation to end of study treatment (Day 27-33)
  This was assessed using the validated questionnaire Nasal Obstruction Symptom Evaluation (NOSE). The total score ranges from 0 to 20, and a higher score indicates more severe nasal obstruction.

OTHER OUTCOMES:
Safety: Frequency and severity of adverse events (AEs), adverse device effects (ADEs), device deficiencies, serious adverse events (SAEs), and serious adverse device effects (SADEs) | From randomisation to end of study i.e., Day 56 (visit window: Day 49 to Day 68)
Safety: Patient-reported addiction score at the follow-up registration (1 question score) | Visit 3 (follow-up registration), i.e., Day 56 (visit window: Day 49 to Day 68)
  The addiction score was designed as a yes/no question.

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Høye, MD, Study Director — Pharma Nordic AS
Locations (7):
- Norway (7):
  - Bjørge Øre-Nese-Hals, Ålesund
  - Haukeland Universitetssykehus, Departments of Otolaryngology and Head and Neck Surgery, Helse Bergen, Bergen
  - Stortorget Øre Nese Hals AS, Hamar
  - Hov Legesenter, Hov
  - Sørlandet Sykehus, Kristiansand, Department for Ear, Nose and Throat, Kristiansand
  - Heiaklinikken Legesenter, Helsehuset Lierskogen, Lierskogen
  - Stavanger Øre-Nese-Hals, Stavanger

IPD SHARING:
Plan to Share IPD: No